CLINICAL TRIAL: NCT04004780
Title: Prevalence of Self-medication for Dental Conditions by Parents for Their Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Faten Salah Abdel-Moniam, Doctor, Cairo University
Other Study IDs: dental self-medication
Record Dates: First submitted 2019-06-27; First posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Self-medication for Dental Conditions
Keywords: Self-medication-drug interactions

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate prevalence of self-medication for dental conditions by parents for their children.

Self-medications practices.

DETAILED DESCRIPTION:
According to the World Health Organization, self-medication is the act of medicating oneself, either on their own initiative or on the advice of a close person, to treat self-recognized conditions or symptoms without supervision by a healthcare professional.

The growth and dissemination of self-medication practice represents a serious global public health issue, with increased risks of adverse drug reactions, non-beneficial drug interactions, drug abuse, and the emergence of drug-resistant pathogens.

Parents are the primary caregivers to whom children report their symptoms. But due to the presence of economic and time constraints, some parents seek the practice of self-medication for their children . However, children have a growing body reacting differently to the drugs (need of dose adjustment, choice of the proper route of administration and the need of taking in consideration the pharmacokinetics and pharmacodynamics particularities of medicines) and therefore the inappropriate and unguided use of medications may lead to fatal complications.

ELIGIBILITY:
Inclusion Criteria:

* Parents of healthy children up to 10 years.
* Parents who accept to participate in the study

Exclusion Criteria:

* Guardians other than parents (child's father or mother).

Ages: 3 Years to 10 Years | Sex: All
Age Groups: Child
Study Population: Parents of healthy children up to 10 years.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
prevalence of self-medication | one year
  Questionnaire (binary or MSQ questions)

SECONDARY OUTCOMES:
self-medication practices | one year
  Questionnaire (binary or MSQ questions)

REFERENCES:
- [Background] • Dentistry, P. (2018). RESEARCH ARTICLE SELF-MEDICATION MEDICATION PRACTICES BY PARENTS IN CHILDREN FOR DENTAL CONDITIONS * Amrita Amrita Nayyar and Anand K. Tavargeri Department of Pediatric and Preventive Dentistry, SDM College of Dental Sciences and Hospital
- [Background] • Paulino, M. R., Clementino, M. A., Santos, H. B. de P., Batista, M. I. H. de M., Carvalho, A. A. T., Nonaka, C. F. W., & Sousa, S. A. de. (2019). Self-Medication for Toothache and its Associated Factors in Children and Adolescents. Pesquisa Brasileira Em Odontopediatria e Clínica Integrada, 19(1), 1-9. https://doi.org/10.4034/pboci.2019.191.3
- [Background] • Santos ANM, Nogueira DRC, Borja-Oliveira CR. Self-medication among participants of an open university of the third age and associated factors. Rev Bras Geriatr Gerontol 2018; 21(4):419-27. https://doi.org/10.1590/1981-22562018021.170204
- [Background] • Bras Odontopediatria Clin Integr 2016; 16(1):229-34. https://doi.org/10.4034/PBOCI.2016.161.24.